CLINICAL TRIAL: NCT05494229
Title: Autologous Whole Blood for Closing Full-thickness Macular Hole
Brief Title: Autologous Blood for Full-thickness Macular Hole
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to complications
Sponsor: Omer Othman Abdullah (Other)
Responsible Party: Sponsor-Investigator, Omer Othman Abdullah, Associate consultant ophthalmologist, Ibinsina Modern Eye and Retina Center
Organization: Ibinsina Modern Eye and Retina Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMER 111
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Ophthalmopathy
Keywords: Full Thickness Macular Hole; Blood Clot; Whole blood; Pars-pana vitrectomy
MeSH Terms: conditions — Eye Diseases; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utilizing autologous whole blood for the full thickness macular hole (Experimental): It is an interventional study by performing pars-plana vitrectomy
  Interventions: Other: Pars-plana vitrectomy

INTERVENTIONS:
Other: Pars-plana vitrectomy — Pars-plana vitrectomy

SUMMARY:
Autologous blood for primary and recurrent holes

DETAILED DESCRIPTION:
Utilizing whole autologous blood for closing both primary and recurrent holes. Here, we apply a drop of the taken whole blood over the hole, and the access blood will be aspirated on the macula with a silicon-tipped active back-flash cannula, to abolish all the possibilities of the fibrinogenic behavior of the whole blood composition, which might cause traction and recurrent hole formation. Therefore, only the hole will be filled with blood. The blood will be taken under completely sterile and aseptic conditions.

The air infusion will be raised after the valve of one of the trocars will be removed, to allow the air current to dry the clot inside the hole rapidly. Then air gas exchange will be performed to allow the clot to remain away from intraocular fluids for one to two weeks and abolish the possibility of the clot being dissolved.

ELIGIBILITY:
Inclusion Criteria:

* Primary and recurrent holes

Exclusion Criteria:

* Lamellar and pseudoholes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Anatomical outcome | The fourth week post-operatively
  OCT

SECONDARY OUTCOMES:
Functional outcome | The fourth week post-operatively.
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Omer Abdullah, M.Sc., Principal Investigator — Ibinsina Modern Eye and Retina Center
Locations (1):
- Omer Othman Abdullah, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No